CLINICAL TRIAL: NCT04694222
Title: Evaluation of Efficacy of LANAP and Adjunctive LLLT Application in the Treatment of Periodontitis: A Randomized Controlled Clinical Study
Brief Title: Use of Laser Assisted New Attachment Procedure and Low Level Laser Therapy for Periodontitis Patients
Acronym: LANAP LLLT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Collaborators: Turkısh Medicines And Medical Devices Agency (Unknown)
Responsible Party: Principal Investigator, Fadime KAYA DADAS, principal investigator, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-TDU-DİŞF-0040
Record Dates: First submitted 2020-12-30; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Periodontitis
Keywords: Laser Assisted New Attachment Procedure; Low Level Laser Therapy; periodontitis; non-surgical periodontal therapy
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: single-blind randomized controlled clinical study
Who Masked: Outcomes Assessor
Masking Description: Clinical measurements were performed by a masked calibrated researcher to provide blindness
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Control Group (Other): scaling and root planning (SRP) was applied.
  Interventions: Device: Nd:YAG laser
- LANAP Group (Active Comparator): After scaling and polishing, three LANAP stages were performed : In the first stage, Nd:YAG laser was applied. In the second stage, full mouth SRP procedure was performed. In the third stage, Nd:YAG laser was applied again.
  Interventions: Device: Nd:YAG laser
- LLLT Group (Active Comparator): after SRP Low Level Laser Therapy was performed using Nd:YAG laser.
  Interventions: Device: Nd:YAG laser
- LANAP+LLLT Group (Active Comparator): after scaling both LANAP and LLLT were applied.
  Interventions: Device: Nd:YAG laser

INTERVENTIONS:
Device: Nd:YAG laser — For LANAP, the fiber optic tip of the Nd:YAG laser (1064 nm) (Fotona Fidelis AT, USA) was used. For LLLT R24 biostimulation handpiece tip (950-μm) Nd:YAG laser (1064 nm) was used.

SUMMARY:
In this study, it is evaluated the effects of laser assisted new attachment procedure (LANAP) and low level laser therapy (LLLT) and on clinical, biochemical and radiographic parameters in addition to non-surgical periodontal treatment (NSPT).

DETAILED DESCRIPTION:
The study was designed as a randomized-controlled, single-blind and parallel design consisting of 80 patients with chronic periodontitis. Study consists of 4 groups, with 20 patients in each group. Group 1 received only NSPT, Group 2 received NSPT+LANAP, Group 3 received NSPT+LLLT, and Group 4 received NSPT+LANAP+LLLT. Clinical measurements of patients and gingival crevicular fluid (GCF) were taken before treatment and after 1 and 3 months. In GCF, interleukin-1beta, interleukin-10 and vascular endothelial growth factor were analyzed. Standard periapical radiographs were taken for radiographic measurements.

In moderate (4-6 mm) and deep pockets (7 mm and above), it was found that all groups treated with laser significantly decrease pocket depth (PD) and clinic attachment level (CAL) compared to Group 1. Group 3 caused significantly less gingival recession than all other groups. There was no statistical difference between the groups in biochemical markers. Radiographic analysis revealed that only Group 2 achieved significant bone filling compared to Group 1.

Bot LANAP and LLLT application in the deep pockets provide an additional contribution to NSPT. It has been found that LLLT administration leads to decrease in PD by creating a minimum recession.

ELIGIBILITY:
Inclusion Criteria:

* periodontitis of periodontal stage II, III, or IV with grades B
* with at least 12 teeth in the mouth and had ≥4 teeth but not all of them in the same quadrant
* with Probing depth of ≥5 mm, Clinical attachment level of ≥4 mm
* radiographic evidence of alveolar bone loss

Exclusion Criteria:

* smoking
* pregnancy and lactation
* using antibiotics in the last 6 months and anti-inflammatory drugs in the last 3rd months,
* having the systemic disease and the use of the drug that will affect the periodontal condition, having restoration of the adjacent tooth to be collected gingival crevicular fluid

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-04-16 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Clinical attachment level gain | Baseline
  The clinical attachment level is determined by measuring the distance from the cemento-enamel junction to the gingival margin and adding the pocket depth to it.
Clinical attachment level gain | 1 month
  The clinical attachment level is determined by measuring the distance from the cemento-enamel junction to the gingival margin and adding the pocket depth to it.
Clinical attachment level gain | 3 month
  The clinical attachment level is determined by measuring the distance from the cemento-enamel junction to the gingival margin and adding the pocket depth to it.

SECONDARY OUTCOMES:
Probing depth | Baseline
  It is determined by measuring the distance from the gingival margin to the pocket base
Probing depth | 1 Month
  It is determined by measuring the distance from the gingival margin to the pocket base
Probing depth | 3 Month
  It is determined by measuring the distance from the gingival margin to the pocket base
Gingival index | Baseline
  For assessing severity of gingivitis, and its location by examining qualitative changes of gingival tissues
Gingival index | 1 Month
  For assessing severity of gingivitis, and its location by examining qualitative changes of gingival tissues
Gingival index | 3 Month
  For assessing severity of gingivitis, and its location by examining qualitative changes of gingival tissues
Plaque index | Baseline
  This index measures the thickness of plaque on gingival one third
Plaque index | 1 Month
  This index measures the thickness of plaque on gingival one third
Plaque index | 3 Month
  This index measures the thickness of plaque on gingival one third
Bleeding on probing | Baseline
  In this index, probing is performed by gently walking around the pocket and bleeding is evaluated. As a result of probing, evaluation is made by looking at the presence or absence of bleeding in the gingiva.
Bleeding on probing | 1 Month
  In this index, probing is performed by gently walking around the pocket and bleeding is evaluated. As a result of probing, evaluation is made by looking at the presence or absence of bleeding in the gingiva.
Bleeding on probing | 3 Month
  In this index, probing is performed by gently walking around the pocket and bleeding is evaluated. As a result of probing, evaluation is made by looking at the presence or absence of bleeding in the gingiva.
Interleukin-1beta | Baseline
  IL-1 is a protein produced mainly by monocytes and macrophages as a polyclonal activator.
Interleukin-1beta | 1 Month
  IL-1 is a protein produced mainly by monocytes and macrophages as a polyclonal activator.
Interleukin-1beta | 3 Month
  IL-1 is a protein produced mainly by monocytes and macrophages as a polyclonal activator.
Interleukin-10 | Baseline
  IL-10 is an 18 kilodalton (KD) cytokine with a wide variety of (pleiotropic) effects.
Interleukin-10 | 1 Month
  IL-10 is an 18 kilodalton (KD) cytokine with a wide variety of (pleiotropic) effects.
Interleukin-10 | 3 Month
  IL-10 is an 18 kilodalton (KD) cytokine with a wide variety of (pleiotropic) effects.
vascular endothelial growth factor (VEGF) | Baseline
  VEGF is a glycoprotein molecule that is a potential stimulator of angiogenesis.
vascular endothelial growth factor (VEGF) | 1 Month
  VEGF is a glycoprotein molecule that is a potential stimulator of angiogenesis.
vascular endothelial growth factor (VEGF) | 3 Month
  VEGF is a glycoprotein molecule that is a potential stimulator of angiogenesis.
Radiographic bone fill | Baseline
  The effects of treatments on bone loss were evaluated by making some measurements on periapical radiography.
Radiographic bone fill | 1 Month
  The effects of treatments on bone loss were evaluated by making some measurements on periapical radiography.
Radiographic bone fill | 3 Month
  The effects of treatments on bone loss were evaluated by making some measurements on periapical radiography.

CONTACTS AND LOCATIONS:
Overall Officials: Serhat Köseoğlu, Study Director — study manager
Locations (1):
- Katip Celebi University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaya Dadas F, Genc Kocaayan S, Saglam M, Dadas OF, Koseoglu S. Evaluating efficacy of laser-assisted new attachment procedure and adjunctive low-level laser therapy in treating periodontitis: A single-blind randomized controlled clinical study. Lasers Med Sci. 2025 Apr 22;40(1):208. doi: 10.1007/s10103-025-04457-0. PMID 40259146

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-11-22): https://cdn.clinicaltrials.gov/large-docs/22/NCT04694222/SAP_000.pdf